CLINICAL TRIAL: NCT03615638
Title: Effectiveness of a Community-based Post-operative Rehabilitation and Fall Prevention Program Following Total Knee Arthroplasty - a Randomized Controlled Trial
Brief Title: Community-based Rehabilitation and Fall Prevention Program After Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Neuroscience Research Australia (Other)
Responsible Party: Principal Investigator, Dr Arnold Wong Yu Lok, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSEARS20171225001
Record Dates: First submitted 2018-07-31; First posted 2018-08-06 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Knee Osteoarthritis; Fall
Keywords: Fall prevention; Total knee arthroplasty; Commnuity-based
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Single-blinded 3-arm randomized controlled trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The orthopedic surgeons, outcomes assessor and statistician will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fall prevention group (Experimental): Fall prevention program
  Interventions: Other: Fall prevention program
- Usual care group (No Intervention): Usual postoperative care
- Asymptomatic control (No Intervention): No intervention

INTERVENTIONS:
Other: Fall prevention program — 12-week fall prevention program (including warm-up, cool-down, education, Tai Chi, and lower limb strengthening)
  Arms: Fall prevention group

SUMMARY:
Knee osteoarthritis (OA) is a common musculoskeletal disorder among older people. Since the prevalence of knee OA increases with age, it is anticipated that the prevalence and burden of knee OA will increase significantly given the aging population.

Total knee arthroplasty (TKA) is used to treat patients with severe knee OA. While TKA has been shown to improve knee pain, function and quality of life of patients with knee OA, up to 50% of patients with post-TKA may suffer from falls within in the first year after TKA. Given that Tai Chi can significantly improve the balance and function of older people, a fall prevention program may improve balance, pain, and function of post-TKA patients.

As such, the current 3-arm randomized controlled trial (RCT) aims to compare the effectiveness of a post-operative community-based fall prevention program in improving knee pain, function and balance of patients with unilateral TKA against a group of TKA patients receiving standard post-operative care, and age- and gender-matched asymptomatic controls over 1 year.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the third most disabling musculoskeletal compliant in the world. Knee OA is the most common type of OA. Since the prevalence of knee OA increases with age, it is anticipated that the prevalence and burden of knee OA will increase significantly given the aging population.

Total knee arthroplasty (TKA) is a surgical intervention for treating patients with severe knee OA. Research has found that TKA reduces knee pain, and improves patient's function and quality of life. However, studies have also found that patients with post-TKA may be more likely to fall as compared to age- and gender-matched asymptomatic counterparts. It is estimated that around 20% to 50% of patients fall within in the first year after TKA. As such, it is essential to improve the balance of post-TKA patients.

Studies have found that Tai Chi can significantly improve the balance and function of older people. Therefore, a fall prevention program aiming at strengthening, proprioception, balance training, and behavioral modification may improve balance, pain, and function of post-TKA patients.

As such, the current 3-arm randomized controlled trial (RCT) aims to compare the effectiveness of a post-operative community-based fall prevention program in improving knee pain, function and balance of patients with unilateral TKA with a group of patients receiving standard post-operative care, and age- and gender-matched asymptomatic controls over 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Participants undergoing TKA for intervention group and usual postoperative care group
* Age- and gender-matched asymptomatic controls without knee pain in the last 12 months.
* Can speak and understand Cantonese/English.

Exclusion Criteria:

* Living in assisted living facilities, requiring nursing care
* Medical 'red flag' conditions
* A history of cancer in the last five years
* Cauda equine syndrome
* Knee fracture
* Auto-immune disease (e.g. rheumatoid arthritis) even if they have OA
* Inflammatory or septic arthritis
* Systemic disease
* Amputation
* History of orthopedic or neurological surgery to the spine, pelvis or hips
* Neurological diseases (e.g. stroke or Parkinson's disease)
* Mini-Mental State Examination score < 24
* Depression subscale score of Depression Anxiety Stress Scales > 21
* Severe comorbidity leading to severe deterioration of quality of life or major healthcare utilization
* Osteochondritis dissecans
* Perthes' disease
* Plica disease
* Baker's cyst

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Chinese version of Knee Injury and Osteoarthritis Outcome Scale | 1 year
  A 42-item questionnaire with 5 subscales to assess pain, symptoms, activities of daily living, sports and recreation function, and knee-related quality of life

SECONDARY OUTCOMES:
11-point numeric pain rating scale | 1 year
  This scale quantify pain on a scale of 0 to 10. Higher the scores, higher the pain intensity
Chinese version Falls Efficacy Scale - International | 1 year
  To examine a person's confidence in avoiding a fall during 16 non-threatening activities of daily living.
Number of post-operative trips/falls | 1 year
  To quantify the number of trips/falls over 1 year after TKA
Chinese version geriatric depression scale | 1 year
  It consists of 15 questions to assess depression in older people
Chinese version Insomnia Severity Index | 1 year
  It assesses sleep problems and related difficulties
Physical Activity Scale for the Elderly | 1 year
  It evaluates leisure, physical, household and work-related activities over the last 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Arnold Wong, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (2):
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Yan Chai Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lo CWT, Brodie MA, Tsang WWN, Yan CH, Lam PL, Chan CM, Lord SR, Wong AYL. Acceptability and feasibility of a community-based strength, balance, and Tai Chi rehabilitation program in improving physical function and balance of patients after total knee arthroplasty: study protocol for a pilot randomized controlled trial. Trials. 2021 Feb 11;22(1):129. doi: 10.1186/s13063-021-05055-5. PMID 33573664